CLINICAL TRIAL: NCT02173431
Title: Mapping Pressure of Human Body to Prevent Bedsores
Brief Title: Recognize High Pressure Areas in Human Body to Prevent Decubitus Ulcers
Acronym: BEDSORES
Status: Withdrawn | Type: Observational
Why Stopped: due to technical issues
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, MD, Assuta Medical Center
Other Study IDs: SCO0414; relation of pressure in gender (Registry Identifier: BMI and pressure mapping)
Record Dates: First submitted 2014-04-10; First posted 2014-06-25 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Pressure Ulcer Stage 1
Keywords: BMI; Pressure; Bedsore
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: None Retained — messure of pressure of patients resting on the buttres with pressure sensors
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- BMI 20 to 24.99: 30 patients
- BMI 25 to 29.99: 30 patients
- BMI 30 to 34.99: 30 patients
- BMI 35 to 39.99: 30 patients
- BMI 40 to 44.99: 30 patients
- BMI 45 to 49.99: 30 patients
- BMI more than 50: 30 patients

SUMMARY:
Prolonged external pressure to the tissue leads to compression, ischemia and development of pressure ulcer.

Underweight seems to be associated with high pressure ulcer risk but the distinct relation between overweight and pressure ulcer development is uncertain.

Bedsores are caused by pressure against the skin that limits blood flow to the skin and nearby tissue.

Others factors related to limited mobility can make the skin vulnerable to damage and contribute to the development of pressure sores. Three primary contributing factors are sustained pressure, friction and shear.

Bedsores are easier to prevent than to treat.

DETAILED DESCRIPTION:
* age
* weight
* high
* BMI
* pressure scanning map
* Alimentary status
* Diseases

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted for elective surgery,
* Patients above 18 y.o.,
* Patient admitted for surgery that required 3 or more days in hospital

Exclusion Criteria:

* Patients under 18
* Patients that require emergency surgery
* Patients that have bedsores before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from 18 y.o. before elective operation will be recruited for the study/ Any patient will be enroled in each group' seven in total according the BMI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Mapping body pressure | up to 6 month
  The patient need to rest above a mattress with sensors for pressure and the data is obtained by an specific software

CONTACTS AND LOCATIONS:
Overall Officials: Sergio G Susmallian, M.D., Principal Investigator — ASSUTA MC
Locations (1):
- ASSUTAMC, Tel Aviv, Israel